CLINICAL TRIAL: NCT05987306
Title: A Self-compassion Focused Intervention for Internalized Weight Bias and Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Carolina University (Other)
Collaborators: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCIRB 23-001492
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single group pre and posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): a standard weight loss and internalized weight bias intervention with self-compassion exercises
  Interventions: Behavioral: Weight loss plus self-compassion

INTERVENTIONS:
Behavioral: Weight loss plus self-compassion — A novel weight loss approach combining a standard weight loss based on the Diabetes Prevention Program and internalized weight bias intervention with self-compassion exercises.

SUMMARY:
The goal of clinical trial is to test a novel weight loss approach combining a standard weight loss and internalized weight bias intervention with self-compassion exercises in overweight adults with moderate to high levels of internalized weight bias. The main question[s] it aims to answer are: 1) Can participants lose significant weight loss and 2) significantly reduce internalized weight bias. Participants will take part in a 12 week novel weight loss approach combining a standard weight loss and internalized weight bias intervention with self-compassion exercises using videoconferencing software.

DETAILED DESCRIPTION:
The goal of clinical trial is to test a novel weight loss approach combining a standard weight loss and internalized weight bias intervention with self-compassion exercises in overweight adults with moderate to high levels of internalized weight bias. The main question[s] it aims to answer are: 1) Can participants lose significant weight loss and 2) significantly reduce internalized weight bias. Participants will take part in a 12-week novel weight loss approach combining a standard weight loss and internalized weight bias intervention with self-compassion exercises using videoconferencing software. The weight loss approach will be modeled after the Diabetes Prevention Program and the approach utilized to reduce internalized weight bias will be Kristen Neff's self-compassion intervention. Each weekly session will utilize Webex videoconferencing software and last approximately 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25, ≥ 18 years old
* Smartphone access
* WBIS score ≥ 4

Exclusion Criteria:

* Type I diabetes, uncontrolled hypertension, cardiovascular event in past year, any major active kidney, liver, cardio, or cerebrovascular disease,
* musculoskeletal problems that would prevent physical activity,
* current weight loss medication or weight loss program,
* history of bariatric surgery,
* pregnant or breastfeeding,
* eating disorder except binge eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Weight (lbs) | 12 weeks
  Change in weight or percent body weight
Weight Bias Internalization Scale | 12 weeks
  Change in internalized weight bias (range 1-7 with higher scores indicating greater internalized weight bias)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Carels, Principal Investigator — East Carolina University
Locations (2):
- United States (2):
  - East Carolina University, Greenville, North Carolina
  - ECU, Dept of Psychology, 104 Rawl, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
I am happy to make data available to qualified researchers.